CLINICAL TRIAL: NCT02155907
Title: Detection of Atrial Fibrillation in Patients With Recent Stroke or TIA: Validity of Automated Loop-recording (R.Test) Compared to Holter Recording and Predictive Value of Short Term Runs of Atrial Fibrillation and SVE for a New Stroke
Brief Title: Atrial Fibrillation Detected by ELR and Holter Recording, a Comparison in Patients With Ischemic Stroke or TIA
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Hospitalsenheden Vest (Other)
Responsible Party: Sponsor
Other Study IDs: Rtest
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2016-06

CONDITIONS: Stroke; Ischaemic Stroke; Atrial Fibrillation; Supra Ventricular Extra Systoles
MeSH Terms: conditions — Stroke; Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Rtest, Atrial fibrillation: Patients with ischemic stroke or TIA within the last week. Sinus rhythm on the surface ECG. Age ≥ 60 years. Given written informed consent

SUMMARY:
Purpose

1. To validate 2 -day loop recording ( R.Test Evolution 4 ) to 2 -day Holter recording (gold standard) for the detection of atrial fibrillation of ≥ 30 seconds duration in a consecutive population of patients with stroke or transient ischemic attack (TIA).
2. To determine whether short run of atrial fibrillation (< 30s ) or the presence of many supraventricular extrasystoles detected on Holter recording, is associated with risk of re-stroke in a consecutive population of patients with stroke or TIA .
3. To test whether a 7-day Loop Recording (R -test) detects more patients with atrial fibrillation than 2 days of Holter recording in a consecutive population of patients with stroke or TIA.

DETAILED DESCRIPTION:
Project title:

Detection of atrial fibrillation in patients with recent stroke or TIA: Validity of automated loop-recording (Rtest) compared to Holter recording and predictive value of short runs of atrial fibrillation and an excess supraventricular extra systoles for a new stroke

Abstract:

Stroke constitutes a major health problem both nationally and globally. Each year 15 million people worldwide are attacked by stroke. In Denmark stroke hits 14.000 people a year and is the third leading cause of death. In this research project, we will examine the heart rate of more than 1,500 patients whom within 1 week has had a blood clot in the brain (ischemic stroke) or have had symptoms of a blood clot in the brain, which has dwindled within 24 hours (TIA). There are no clear international or national guidelines regarding the optimal way to detect atrial fibrillation in stroke and TIA patients, though atrial fibrillation is known to increase fivefold the risk of stroke. Holter recording with two days electrocardiogram is considered as the golden standard for investigation of heart rhythm disturbances and is offered at Department of Neurology in Holstebro, where we recruit patients. Holter recording is a resource-intensive procedure in data analysis. Project patients will be mounted with a 2- day Holter and Rtest for either 2 or 7 days. The Rtest is a loop recorder and a new device on the market that continuously monitor and opposite a Holter recorder, automatically analyses heart rhythm. The validity of the Rtest with regard to detect atrial fibrillation compared to Holter is unknown and is what we which to clarify. Additionally we use the 2-day Holter recordings to test whether short-term rhythm disorders as atrial fibrillation <30 seconds, and/or many extra heartbeats (supraventricular extra systoles) increases the risk of stroke recurrence. Patients will be followed in the Danish Stroke Register. If an increased risk is found, these gray area patients who are currently not offered anticoagulant therapy, may prove to have treatment indication. If the study shows that loop recording can replace Holter recording it will mean an economic gain. The study is expected to contribute substantial evidence for the future treatment of stroke and TIA patients.Stroke constitutes a major health problem both nationally and globally. Each year 15 million people worldwide are attacked by stroke. In Denmark stroke hits 14.000 people a year and is the third leading cause of death. In this research project, we will examine the heart rate of more than 1,500 patients whom within 1 week has had a blood clot in the brain (ischemic stroke) or have had symptoms of a blood clot in the brain, which has dwindled within 24 hours (TIA). There are no clear international or national guidelines regarding the optimal way to detect atrial fibrillation in stroke and TIA patients, though atrial fibrillation is known to increase fivefold the risk of stroke. Holter recording with two days electrocardiogram is considered as the golden standard for investigation of heart rhythm disturbances and is offered at Department of Neurology in Holstebro, where we recruit patients. Holter recording is a resource-intensive procedure in data analysis. Project patients will be mounted with a 2- day Holter and Rtest for either 2 or 7 days. The Rtest is a loop recorder and a new device on the market that continuously monitor and opposite a Holter recorder, automatically analyses heart rhythm. The validity of the Rtest with regard to detect atrial fibrillation compared to Holter is unknown and is what we which to clarify. Additionally we use the 2-day Holter recordings to test whether short-term rhythm disorders as atrial fibrillation <30 seconds, and/or many extra heartbeats (supraventricular extra systoles) increases the risk of stroke recurrence. Patients will be followed in the Danish Stroke Register. If an increased risk is found, these gray area patients who are currently not offered anticoagulant therapy, may prove to have treatment indication. If the study shows that loop recording can replace Holter recording it will mean an economic gain. The study is expected to contribute substantial evidence for the future treatment of stroke and TIA patients.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic stroke or TIA within the last week. Sinus rhythm on the surface ECG. Age ≥ 60 years. Given written informed consent.

Exclusion Criteria:

* AF detected during hospitalization or earlier. Dementia or suspected non-compliance. Known cancer except c prostate with normal PSA, or basal cell carcinoma. Pacemaker or a defibrillator implanted

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke and TCI patients admitted to the Regional Hospital Holstebro
Sampling Method: Non-Probability Sample
Enrollment: 1507 (Actual)
Dates: Start 2013-06-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of restroke | 1 year
  Do short runs of atrial fibrillation < 30 seconds and/or many supraventricular extra systoles increase the risk of restroke?

SECONDARY OUTCOMES:
Validity of looprecordong (R. Test 4 Evolution) compared to Holter recording | 2-7 days pr. patient
  Patients will be monitored with both an Holter recorder an a Rtest at the same time in respectively 2 and 2-7 days

CONTACTS AND LOCATIONS:
Overall Officials: Michala H Sejr, MD, Principal Investigator — University of Aarhus
Locations (1):
- Regional Hospital of Herning, Cardiovascular Research Unit, Medical Department, Herning, Jutland, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sejr MH, May O, Damgaard D, Sandal BF, Nielsen JC. External continuous ECG versus loop recording for atrial fibrillation detection in patients who had a stroke. Heart. 2019 Jun;105(11):848-854. doi: 10.1136/heartjnl-2018-314186. Epub 2019 Mar 21. PMID 30898849